CLINICAL TRIAL: NCT06290752
Title: Associate Chief Physician
Brief Title: Determining the Learning Curve for Ultrasound-guided Caudal Epidural Block
Status: Recruiting | Type: Observational
Sponsor: The Fourth Affiliated Hospital of Zhejiang University School of Medicine (Other)
Responsible Party: Sponsor
Other Study IDs: KY-2024-030
Record Dates: First submitted 2024-02-26; First posted 2024-03-04 (Actual); Last update posted 2024-03-12 (Actual); Status verified 2024-03

CONDITIONS: Anesthesia

STUDY DESIGN:
Observational Model: Ecologic or Community | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
mastering ultrasound-guided sacral canal block entails traversing a multifaceted learning curve characterized by anatomical intricacies, technical challenges, and patient variability. Through systematic education, deliberate practice, and clinical experience, clinicians can ascend this learning curve and harness the full potential of this innovative technique in pain management. As the landscape of regional anesthesia continues to evolve, a commitment to ongoing learning and proficiency attainment is paramount for delivering safe, effective, and patient-centered care.

ELIGIBILITY:
Inclusion Criteria:

* Residential training students in the first -third grade

Exclusion Criteria:

* No-resident trainees

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Residential trainee
Sampling Method: Non-Probability Sample
Enrollment: 6 (Estimated)
Dates: Start 2024-03-01 (Estimated); Primary Completion 2024-11-30 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
operation time | 15 minutes
  Operating time of students from starting scan to nerve block completion

CONTACTS AND LOCATIONS:
Overall Officials: Dongmei Ma, Study Chair — 浙江大学医学院附属第四医院
Locations (1):
- Dongmei Ma, Yiwu, Zhejiang, China

IPD SHARING:
Plan to Share IPD: No